CLINICAL TRIAL: NCT04030611
Title: Assessment the Sensitivity of Traditional Chinese Medical Diagnostic Tools for Diabetic retinopathy-a Pilot Study
Brief Title: The Sensitivity of Traditional Chinese Medical Diagnostic Tools for Diabetic Retinopathy Diabetic retinopathy-a Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH107-REC3--116
Record Dates: First submitted 2019-07-18; First posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetic retinopathy, traditional Chinese medicine(TCM), Diagnositic tools, sensitivity, Blood stasis
MeSH Terms: conditions — Diabetic Retinopathy; Hypersensitivity | interventions — Pulse Wave Analysis; Microscopic Angioscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: Participants in the type 2 DM group were diagnosed with DM based on criteria recommended by the American Diabetes Association and required to have a fasting plasma glucose of ≥7mmol/L or an HbA1c of ≥6.5%, as measured on 2 separate occasions.
  Interventions: Diagnostic Test: tongue diagnosis system
- diabetic retinopahty group: Participants in th ediabetic retinopahty group group were diagnosed according to the International Clinical Diabetic Retinopathy and Diabetic Macular Edema Disease Severity Scales.
  Interventions: Diagnostic Test: tongue diagnosis system

INTERVENTIONS:
Diagnostic Test: tongue diagnosis system — This study apply TCM diagnostic tools for clinical diseases, providing objective diagnostic data for evaluation to assess the association of blood stasis and DR.
  Other Names: pulse wave analysis; body constitution questionnaires; nailfold capillaroscopy

SUMMARY:
Diabetic retinopathy (DR) is the leading cause of impaired visual function and blindness in adults. The fundus photographs were examined to detect DR. The DR severity was graded non-proliferative diabetic retinopathy (NPDR) and proliferative diabetic retinopathy (PDR) according to the International Clinical Diabetic Retinopathy and Diabetic Macular Edema Disease Severity Scales. The pathogenesis of DR is complex and not fully understood, and platelet aggregation, microvascular damage, microvascular enlargement, leakage, hemorrhage, or obstruction, resulting in retinal hypoxia and retinal neovascularization. Traditional Chinese medicine (TCM) diagnostic tools are non-invasive and convenient. This study apply TCM diagnostic tools for clinical diseases, providing objective diagnostic data for evaluation to assess the association of blood stasis and DR. Furtherly we would evaluate the sensitivity and specificity of TCM diagnostic tools.

This study is a prospective cross-sectional study. We enroll participants form the department of Chinese medicine, China Medical University Hospital. In total, 100 participants , composed of 50 of type 2 diabetes and 50 of diabetic retinopathy, whom previously had a retinal examination. We apply tongue diagnosis system, pulse wave analysis, body constitution questionnaires, and nailfold capillaroscopy to assess the differences of TCM diagnosis in DR.

This study aims to identify the clinical symptoms of DR with TCM diagnostic tools and investigate the pattern difference and treatment for DR. Furtherly, we could design a clinical trial with improving blood circulation to treat or prevent DR, and improve the health status and quality of life in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* type 2 DM group were diagnosed with DM based on criteria recommended by the American Diabetes Association and required to have a fasting plasma glucose of ≥7mmol/L or an HbA1c of ≥6.5%, as measured on 2 separate occasions.

Exclusion Criteria:

* cancer, active liver disease, current pregnancy, active infection, and cerebrovascular disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants in this prospective cross-sectional study were recruited from the outpatient clinic of endocrinology in China Medical University Hospital, Taichung, Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-10-10 (Estimated)

PRIMARY OUTCOMES:
Automatic tongue diagnosis | 12 months
  We observe the tongue features of blood stasis, such as bluish tongue, petechiae, and engorged sublingual vessels, and compare the relationship between diabetic retinopathy and blood stasis.
body constitution questionnaire | 12 months
  We observe the body constitution questionnaires, such as yi deficiency, yang deficiency and phlegm-stasis, and compare the relationship between diabetic retinopathy and blood stasis.
Nailfold videocapillaroscopy (NVC) | 12 months
  We evaluate the capillary density, length, morphology, distribution, presence of enlarged loops or hemorrhages, and blood flow. NVC score was used to quantitate the aforementioned characteristics.
pulse examinatin | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No